CLINICAL TRIAL: NCT01290692
Title: Phase 2 Study To Test The Safety and Efficacy of TVI-Brain-1 As A Treatment For Recurrent Grade IV Glioma
Brief Title: Study To Test the Safety and Efficacy of TVI-Brain-1 As A Treatment for Recurrent Grade IV Glioma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: TVAX Biomedical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TVI-AST-005
Record Dates: First submitted 2011-02-03; First posted 2011-02-07 (Estimated); Results first posted 2023-06-29 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Grade IV Glioma; Grade IV Astrocytoma; Glioblastoma Multiforme
Keywords: Brain Neoplasms; Central Nervous System Neoplasms; Brain Diseases; Neoplasms; Nervous System Neoplasms; Glioblastoma; Astrocytoma; Nervous System Diseases; Central Nervous System Diseases; Glioma; Recurrent astrocytoma; Recurrent glioma; Cancer vaccine; Immunotherapy; Killer T cells; Activated T cells; GM-CSF; Activated lymphocytes
MeSH Terms: conditions — Glioblastoma; Brain Neoplasms; Central Nervous System Neoplasms; Brain Diseases; Neoplasms; Nervous System Neoplasms; Astrocytoma; Nervous System Diseases; Central Nervous System Diseases; Glioma | interventions — Cancer Vaccines; Adjuvants, Immunologic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TVI-Brain-1 (Experimental): All patients will receive the full TVI-Brain-1 treatment.
  Interventions: Biological: TVI-Brain-1

INTERVENTIONS:
Biological: TVI-Brain-1 — Following surgery, tumor tissue is used to generate a cancer vaccine. Patients are vaccinated with neutralized cells to initiate an immune response. Following vaccinations, the patient's white blood cells are collected, the white blood cells are stimulated and expanded, and are then reinfused into the patient's blood.
  Other Names: Cancer vaccine plus immune adjuvant plus activated WBC

SUMMARY:
TVI-Brain-1 is an experimental treatment that takes advantage of the fact that your body can produce immune cells, called 'killer' white blood cells that have the ability to kill large numbers of the cancer cells that are present in your body. TVI-Brain-1 is designed to generate large numbers of those 'killer' white blood cells and to deliver those cells into your body so that they can kill your cancer cells.

DETAILED DESCRIPTION:
The TVI-Brain-1 treatment involves several steps. First, the patient's cancer will be surgically removed to provide cells for the vaccine. Second, the patient will be vaccinated with the vaccine formulation. Third, the patient's blood will be filtered for killer T cell precursors which will then be cultured and stimulated to reach a higher (killer) activity level. Fourth, the activated cells will be infused into the patient's bloodstream so that they will be able to attack the cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* Informed consent
* Diagnosis of grade IV glioma with progression following standard treatment.
* Must be able to tolerate surgery to provide tumor tissue for vaccine.
* Must be able to produce viable vaccine from tumor tissue.
* Karnofsky Performance Status must be 70 or greater.
* Negative HIV test.
* Negative for hepatitis B and C virus.
* Respiratory reserve must be reasonable.
* Sufficient renal function.
* Satisfactory blood counts.
* Negative pregnancy test for women of childbearing potential.

Exclusion Criteria:

* Surgically removed cancer reveals that it is not grade IV glioma.
* Concomitant life-threatening disease.
* Active autoimmune disease.
* Currently receiving chemotherapy or biological therapy for the treatment of cancer.
* Currently receiving immunosuppressive drugs for any reason.
* Prior treatment with Avastin or other anti-angiogenesis treatment within 6 months.
* Prior treatment with Gliadel wafers.
* Corticosteroids beyond peri-operative period.
* Psychological, familial, sociological or geographical conditions that do not permit adequate medical follow-up and compliance with the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2011-06; Primary Completion 2013-12 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary Wood, Ph.D., Study Chair — Sponsor GmbH
Locations (4):
- United States (4):
  - Saint Luke's Hospital, Kansas City, Missouri
  - Washington University, St Louis, Missouri
  - Baylor University Medical Center, Dallas, Texas
  - Aurora BayCare Medical Center, Green Bay, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sloan AE, Dansey R, Zamorano L, Barger G, Hamm C, Diaz F, Baynes R, Wood G. Adoptive immunotherapy in patients with recurrent malignant glioma: preliminary results of using autologous whole-tumor vaccine plus granulocyte-macrophage colony-stimulating factor and adoptive transfer of anti-CD3-activated lymphocytes. Neurosurg Focus. 2000 Dec 15;9(6):e9. doi: 10.3171/foc.2000.9.6.10. PMID 16817692
- See also: Sponsor website — http://www.tvaxbiomedical.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment was prematurely closed to allow a change in protocol design based on clinical findings from the small study. The data justified change in protocol design (study #008) to treat subjects with minimal residual disease and healthy immune system.
Period: Overall Study
Arm/Group | TVI-Brain-1
Started | 14
Completed | 7
Not Completed | 7
Not completed — Lack of sufficient efficacy as patients were immunocompromised | 7

BASELINE CHARACTERISTICS:
Arm/Group | TVI-Brain-1
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 13
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Progression of Disease
Description: To assess the efficacy of TVI-Brain-1 on patients to evaluate progression free survival. MRI data is used to evaluate tumor progression; success is defined if a patient is still alive and has < 25 % increase in Tumor volume in MRI collected at 6 month timepoint.
Time Frame: 6-months
Measure: Count of Participants; unit: Participants
Arm/Group | TVI-Brain-1
Number analyzed (Participants) | 14
Participants | 14

2. Secondary Outcome: Overall Survival
Description: All patients will be followed until death or the end of the study to measure overall survival.
Time Frame: 32 months
Measure: Count of Participants; unit: Participants
Arm/Group | TVI-Brain-1
Number analyzed (Participants) | 14
Participants | 0

3. Secondary Outcome: Number of Participants With Treatment-related Adverse Events as Assessed by CTCAE v4.0
Description: Toxicity will be assessed throughout the study by recording clinical symptoms, performing physical examinations, measuring vital signs and performing clinical laboratory tests, including complete blood counts and differentials, blood chemistries and autoimmune profiles.
Time Frame: 12 weeks
Population: Toxicity was assessed throughout the study by recording clinical symptoms, physical examinations, vital signs, clinical laboratory tests, including blood counts and differentials, blood chemistries and autoimmune profiles. Patients were monitored for toxicities during the study and for one month following removal from the study for any reason.
Measure: Count of Participants; unit: Participants
Arm/Group | TVI-Brain-1
Number analyzed (Participants) | 14
Participants | 14

4. Secondary Outcome: Time to Progression of Tumor Per MRI
Description: Time to progression is defined date of evidence of increase in tumor volume as evaluated by review and analysis of imaging, using MacDonald Criteria in review of serial MRI's taken at specific timepoints
Time Frame: 32-months
Population: MRI data not collected
Arm/Group | TVI-Brain-1
Number analyzed (Participants) | 0

5. Secondary Outcome: Objective Response Rate
Description: Time to progression is defined as assessed by neurologists and radiologists evaluation of time to worsening of patient's neurological status and/or increase in tumor volume measurements as evaluated by review and analysis of serial physical exams and MRI's taken at specific timepoints
Time Frame: 32-months
Population: MRI data not collected nor analyzed
Arm/Group | TVI-Brain-1
Number analyzed (Participants) | 0

6. Secondary Outcome: Delayed-type Hypersensitivity (DTH) Skin Testing
Description: Skin Test using attenuated autologous cancer cells will be performed to assess the immunogenicity of the Subject's cancer.
  Evidence of a Resulting wheal or flare reaction from sub-cutanous injection of test will be evaluated in each patient
Time Frame: 48 hours
Measure: Count of Participants; unit: Participants
Arm/Group | TVI-Brain-1
Number analyzed (Participants) | 14
Participants | 14

7. Secondary Outcome: Quality of Life as Measured by FACT-Br Tool Score
Description: Quality of life data using the FACT-Br score tabulation from responses on validated tool
Time Frame: 32 months
Population: QOL tool data was not collected
Arm/Group | TVI-Brain-1
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 32 months
Description: Adverse events were collected at all clinic visits through evaluation of blood chemistry and hematology labs, vital sign measurements, physical exams, and direct patient questioning.
Arm/Group | TVI-Brain-1
All-Cause Mortality (participants affected / at risk) | 14/14
Serious Adverse Events (participants affected / at risk) | 9/14
Other Adverse Events (participants affected / at risk) | 5/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TVI-Brain-1 (N=14)
Fever and Chills (Immune system disorders) | 3 (3)
Urinary Tract Infection (Renal and urinary disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Hemiparesis (Musculoskeletal and connective tissue disorders) | 1 (1)
Hemisensory Neglect (Nervous system disorders) | 1 (1)
Paresthesia (Nervous system disorders) | 1 (1)
Seizures (Nervous system disorders) | 3 (3)
disorientation (Nervous system disorders) | 1 (1)
Pulmonary Edema (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TVI-Brain-1 (N=14)
Tachycardia (Cardiac disorders) | 1 (1) — Mild AE
Nausea (Gastrointestinal disorders) | 1 (2) — Mild AE
Chills (General disorders) | 3 (6) — Mild AE
Redness at injection sites (General disorders) | 1 (1) — Mild AE
Fever (General disorders) | 2 (5) — Mild AE
Generalized Aching (General disorders) | 1 (1) — Mild AE
Infusion Site irritation/pain (General disorders) | 1 (1) — Mild AE
Rigors (General disorders) | 1 (1) — Mild AE
Calcium Low (Investigations) | 1 (1) — Mild AE
Hypocalcemia (Metabolism and nutrition disorders) | 1 (3) — Mild AE
Hypokalemia (Metabolism and nutrition disorders) | 2 (5) — Mild AE
Hypomagnesae (Metabolism and nutrition disorders) | 1 (2) — Mild AE
Vomiting (Gastrointestinal disorders) | 1 (1) — Moderate AE
Chills (General disorders) | 2 (2) — Moderate AE
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) — Moderate AE
Hypokalemia (Metabolism and nutrition disorders) | 1 (2) — Moderate AE

LIMITATIONS AND CAVEATS:
Recruitment was stopped to allow a change in protocol design. Some positive clinical effects were observed but this study design treated Subjects whose cancers have progressed following surgery, radiotherapy, and temozolomide chemotherapy and therefore have immune systems that are too compromised to allow maximal benefit from the use of TVI-Brain-1. Study #008 is changed to treat newly diagnosed Subjects with healthy immune systems and minimal residual disease.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No